CLINICAL TRIAL: NCT03483493
Title: Therapist-guided, Parent-assisted Remote Digital Behavioural Intervention for Tics in Children and Adolescents With Tourette Syndrome: an Internal Pilot Study and Single-blind Randomised Controlled Trial
Brief Title: Online Remote Behavioural Intervention for Tics (ORBIT)
Acronym: ORBIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottinghamshire Healthcare NHS Trust (Other Government)
Collaborators: University College, London (Other); Karolinska Institutet (Other); National Institute for Health Research, United Kingdom (Other Government); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hollis201117
Record Dates: First submitted 2018-03-12; First posted 2018-03-30 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Tic Disorders; Tourette Syndrome
Keywords: Tic disorders; Tourette Syndrome; Online delivered therapy
MeSH Terms: conditions — Tic Disorders; Tourette Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure Response Prevention for tics (Experimental): 10-weeks, online delivered, therapist supported exposure response prevention (ERP) therapy for tics
  Interventions: Behavioral: Exposure Response Prevention for tics
- Active Control (Psychoeducation) (Active Comparator): 10-weeks, online delivered, therapist supported psychoeducation for tics
  Interventions: Other: Psychoeducation for tics

INTERVENTIONS:
Behavioral: Exposure Response Prevention for tics — The intervention consists of evidence-based interventions adapted from previously published treatment manuals on Exposure and Response Prevention (ERP) and established behavioural intervention for tics protocols. Each of the 10 modules includes age-appropriate texts, animations and exercises. Prticipants are instructed to practice suppressing their tics, this is known as 'response prevention'. Then, with the help of their parent/carer, the participant is instructed to provoke premonitory urges (the urge to tic often felt before the tic is expressed) and try to supress the need to express/demonstrate the tic, this known as 'exposure'.
  Arms: Exposure Response Prevention for tics
Other: Psychoeducation for tics — The comparator intervention reviews the definition of tics, natural history, common presentations, prevalence, aetiology, risks and protective factors and strategies for describing tics to other people etc. Problem-solving and development of expertise in tic disorders is emphasised. The intervention includes strategies for promoting positive behaviours which will be rewarded by a parent as a parallel element to the tic control practice in the behavioural therapy arm. There is no information on tic control within the management package.
  Arms: Active Control (Psychoeducation)

SUMMARY:
Online Remote Behavioural Intervention for Tics (ORBIT).

Primary objective: to evaluate the clinical effectiveness of BiP Tic, a therapist-guided, parent-assisted, internet-based behavioural therapy intervention for tics in young people, compared with usual care plus online education.

Secondary objectives include 1) optimising the design of the intervention, 2) undertaking an internal pilot, 3) evaluating cost effectiveness and 4) longer term impact, and 5) identifying barriers to implementation.

DETAILED DESCRIPTION:
The ORBIT (Online Remote Behavioural Intervention for Tics) trial is comparing the effectiveness of two treatments delivered online for children and young people with Tourette Syndrome or Chronic Tic Disorder. Families in England with a child/young person (aged 9-17 years) who experiences tics are being asked to take part. Interested families undergo a telephone screen with a researcher and then asked to complete an online questionnaire. They then attend a screening appointment at either Great Ormond Street Hospital (London) or Queen's Medical Centre (Nottingham).

Families that are eligible and want to take part are randomly allocated to one of two treatments. One treatment uses behavioural therapy (BT), the other involves psychoeducation. Both treatments last for 10-weeks and involve completing online chapters (for the parent and child) with the support of a therapist, there are also some tasks to complete offline. After finishing the treatment, families are asked to complete more questionnaires (at 3, 6, 12 and 18 months after starting the treatment). A smaller sample of families and healthcare professionals are also interviewed about their experience of participation. The study is looking to see if the online delivered treatment may be effective at helping children and young people manage their tics. The study is also exploring whether the online programme is acceptable to families, identifying any problems in getting families to take part/complete the programme and also healthcare professionals' views about the programme. It is important to research online therapy for tics because, at the moment, many people with tics do not get any therapy because there are not enough trained tic therapists. If online delivered treatment is effective, this may mean more children and young people could access tic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 9 to 17: patient confirmed through screening.
2. Suspected or confirmed Tourette syndrome/ chronic tic disorder:

   - Including Moderate/severe tics: Score >15 on the Yale Global Tic Severity Scale (YGTSS) Total Tic Severity Score (TTSS); TTSS score>10 if motor or vocal tics only: researcher confirms at screening appointment
3. Competent to provide written, informed consent (parental consent for child aged <16): researcher confirms at screening appointment.
4. Broadband internet access and regular PC/ laptop/Mac user, with mobile phone SMS: patient confirmed through screening.

Exclusion Criteria:

1. Previous structured behavioural intervention for tics e.g. HRT/CBIT or exposure and response prevention within last 12 months: Patient confirmed through screening.
2. Change to medication for tics (start or stop tic medication) within the previous 2 months: Patient confirmed through screening and subsequent medication/interventions commenced throughout out the trial are recorded at each time point for analysis.
3. Diagnoses of alcohol/substance dependence, psychosis, suicidality, or anorexia nervosa: Confirmed through parent DAWBA. DAWBAs that score people as being likely to have these conditions will be second reviewed by the CI (who is a medical expert) to ascertain that they should definitely be excluded from the trial. If the child is considered at immediate risk of suicide, the research team will inform the GP or usual treating clinician.
4. Moderate/severe intellectual disability: Confirmed through qualitative judgement of the assessor at the telephone screen (and confirmed at baseline through CAIDS-Q) through questions relating to type of school the child attends and previous diagnoses.
5. Immediate risk to self or others: Confirmed through screening questions and DAWBA. The participants GP will be informed of this.
6. Parent or child not able to speak or read/write English: Patient confirmed through screening by the assessor.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Assessing change in tics in participants using the Yale Global Tic Severity Scale - Total Tic score | Baseline, 3, 6, 12 and 18 months
  Investigator administered semi structured symptom checklist of 46 tic disorder symptoms. The Total Tic Score is derived by adding the Total Motor Tic Score and the Total Phonic Tic Score

SECONDARY OUTCOMES:
Assessing change in tics in participants using the Parent Tic Questionnaire | Baseline, 5wks, 3mths, 6mths, 12mths & 18 months
  Self administered questionnaire to collect the number, frequency and intensity of 14 common motor and 14 common vocal tics
Assessing change in symptom severity/improvement in participants using the Clinical Global Impressions Scale. | 3, 6, 12 & 18 months
  Clinician determined measure that summarises the patient's history, symptoms, behaviours and psychosocial circumstances
Assessing change in tic impairment in participants using the Yale Global Tic Severity Scale Impairment Scale (assessing change) | Baseline, 3, 6, 12 & 18 months
  This forms part of the YGTSS but focuses on distress and impairment experienced in the individuals life
Assessing change in global functioning in participants using the Children's Global Assessment Scale | Baseline, 3, 6, 12 & 18 months
  A measure of psychiatric disturbance integrating psychological, social and academic functioning
Assessing change in general functioning in participants using the Strengths and Difficulties Questionnaire | Baseline, 3, 6, 12 & 18 months
  Self-report, parent completed questionnaire measuring behavioural and emotional difficulties in children. The baseline SDQ is completed as part of a screening tool "DAWBA".
Assessing change in mood in participants using the Mood and Feelings Questionnaire | Baseline, 1, 3, 6, 12 & 18 months
  Child completed, self-report questionnaire collecting information on depressive symptoms
Assessing change in anxiety in participants using the Spence Child Anxiety Scale | Baseline, 3, 6, 12 & 18 months
  Self-report child completed questionnaire evaluating symptoms of separation anxiety, social phobia, obsessive-compulsive disorder, pain, agoraphobia, generalised anxiety and fear of physical injury
Assessing change in quality of life in participants using the Child Health Utility 9D | Baseline, 3, 6,12,18 months
  Self-report parent and child completed quality of life measure
Assessing change in tic-related quality of life in participants using the Child and Adolescent Gilles de la Tourette Syndrome | Baseline, 3, 6, 12 & 18 months
  A disease specific measure of health related quality of life for children and adolescents with Tourette Syndrome. There are two version, one for children aged 6-12 years and a second for young people aged 3-8 years
Assessing participants change in use of services using the Modified Client Service Receipt Inventory | Baseline, 3, 6, 12 & 18 months
  A questionnaire to collect information on services received, service related issues, school attendance and family income
Assessing change in side effects in participants using the Adverse events/side effects | Baseline, 1, 3, 6, 12 & 18 months
  A 17 item scale of common side effects
Assessing participants perception of treatment credibility using a specifically created 'treatment credibility' questionnaire | 3 weeks
  A two item questionnaire to assess how well the treatment suits children, according to the perception of the 1) parent/carer and 2) child/young person
Assessing participants perception of treatment satisfaction using a specifically created 'treatment satisfaction' questionnaire | 3 months
  A 7 item scale questionnaire developed for the study to assess treatment satisfaction from the perception of the 1) parent/carer and 2) child/young person
Assessing participants perception of their need for further treatment using a specifically created 'Need for further treatment' questionnaire | 3 months
  A single item questionnaire asking if the child or young person requires more treatment for their tics from the perception of the 1) parent/carer and 2) child/young
Assessing participants change of use of other medication/interventions using a specifically created 'Concomitant interventions' questionnaire | Baseline, 3, 6, 12 & 18 months
  Assessment of any other treatment or interventions the child or young person is accessing during the study
Describing sample characteristics using Development and Wellbeing Assessment (DAWBA) at screening/baseline | Screening/Baseline
  The DAWBA is a package of interviews and questionnaires completed by parents and teachers and designed to generate ICD-10 and DSM-IV / DSM-5 psychiatric diagnoses for children and young people.
Determining presence of an intellectual disability at screening/baseline using the Child and Adolescent Intellectual Disability Screening Questionnaire (CAIDS-Q) | Screening/Baseline
  A 7-item questionnaire to determine the presence of intellectual disability at screening/baseline, completed by the parent/
Understanding the characteristics of the sample a specifically created demographics questionnaire at screening/baseline | Screening/Baseline
  Parent completed questionnaire asking about the child's age, gender, ethnicity, parental education/ occupation, list of the child's current diagnoses and interventions (including medications) and GP and school details.
Determining the for presence of Autism Spectrum Disorder using the Social Communication Questionnaire (SCQ) at screening/baseline | Screening/Baseline
  A 40 item, parent-report questionnaire asking about characteristic autistic behaviour at the age of 4 to 5 years and currently.
Assessing Premonitory urges for tics using the Premonitory Urge for Tics Scale (PUTS) at screening/baseline | Screening/Baseline
  A self-report instrument specifically designed to measure the current frequency of different types of premonitory urges in patients with tic disorders
Assessing ADHD symptoms using the Swanson, Nolan, and Pelham Rating Scale (SNAP-IV) at screening/baseline | Screening/Baseline
  A parent completed 26-item behavioural rating scale that employs the core symptoms of ADHD and oppositional defiance disorder (ODD) as defined by the Diagnostic and Statistical Manual of Mental Disorders.

OTHER OUTCOMES:
To assess the process evaluation of the interventions qualitative interviews will be conducted | 3months
  A sub-sample of participants will be as asked to participate in qualitative interviews as part of a process evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Hollis, MD, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Nottinghamshire Healthcare NHS Foundation Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data are available for use by researchers with a sound research idea from priment@ucl.ac.uk
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available beginning 3 months and ending 5 years after the specified trial outcome paper(s) is/are published.

REFERENCES:
- [Result] Hollis C, Hall CL, Jones R, Marston L, Novere ML, Hunter R, Brown BJ, Sanderson C, Andren P, Bennett SD, Chamberlain LR, Davies EB, Evans A, Kouzoupi N, McKenzie C, Heyman I, Khan K, Kilgariff J, Glazebrook C, Mataix-Cols D, Murphy T, Serlachius E, Murray E. Therapist-supported online remote behavioural intervention for tics in children and adolescents in England (ORBIT): a multicentre, parallel group, single-blind, randomised controlled trial. Lancet Psychiatry. 2021 Oct;8(10):871-882. doi: 10.1016/S2215-0366(21)00235-2. Epub 2021 Sep 1. PMID 34480868
- [Derived] Hall CL, Le Novere M, Murphy T, McNally E, Hollis C, Hunter R. Healthcare utilisation and costs associated with poor access to diagnosis and treatment for children and young people with tic disorders. BMJ Ment Health. 2024 Nov 7;27(1):e301241. doi: 10.1136/bmjment-2024-301241. PMID 39515845
- [Derived] Hollis C, Hall CL, Khan K, Le Novere M, Marston L, Jones R, Hunter R, Brown BJ, Sanderson C, Andren P, Bennett SD, Chamberlain LR, Davies EB, Evans A, Kouzoupi N, McKenzie C, Heyman I, Kilgariff J, Glazebrook C, Mataix-Cols D, Serlachius E, Murray E, Murphy T. Online remote behavioural intervention for tics in 9- to 17-year-olds: the ORBIT RCT with embedded process and economic evaluation. Health Technol Assess. 2023 Oct;27(18):1-120. doi: 10.3310/CPMS3211. PMID 37924247
- [Derived] Hollis C, Hall CL, Khan K, Jones R, Marston L, Le Novere M, Hunter R, Andren P, Bennett SD, Brown BJ, Chamberlain LR, Davies EB, Evans A, Kouzoupi N, McKenzie C, Sanderson C, Heyman I, Kilgariff J, Glazebrook C, Mataix-Cols D, Serlachius E, Murray E, Murphy T. Long-term clinical and cost-effectiveness of a therapist-supported online remote behavioural intervention for tics in children and adolescents: extended 12- and 18-month follow-up of a single-blind randomised controlled trial. J Child Psychol Psychiatry. 2023 Jun;64(6):941-951. doi: 10.1111/jcpp.13756. Epub 2023 Jan 17. PMID 36649686
- [Derived] Hall CL, Marston L, Khan K, Brown BJ, Sanderson C, Andren P, Bennett S, Heyman I, Mataix-Cols D, Serlachius E, Hollis C, Murphy T. The COVID-19 pandemic and its impact on tic symptoms in children and young people: a prospective cohort study. Child Psychiatry Hum Dev. 2023 Dec;54(6):1499-1509. doi: 10.1007/s10578-022-01348-1. Epub 2022 Apr 13. PMID 35416566
- [Derived] Hall CL, Sanderson C, Brown BJ, Andren P, Bennett S, Chamberlain LR, Davies EB, Khan K, Kouzoupi N, Mataix-Cols D, McKenzie C, Murphy T, Townsend M, Hollis C, Murray E. Opportunities and challenges of delivering digital clinical trials: lessons learned from a randomised controlled trial of an online behavioural intervention for children and young people. Trials. 2020 Dec 9;21(1):1011. doi: 10.1186/s13063-020-04902-1. PMID 33298127
- [Derived] Khan K, Hollis C, Hall CL, Davies EB, Mataix-Cols D, Andren P, Murphy T, Brown BJ, Murray E, Glazebrook C. Protocol for the Process Evaluation of the Online Remote Behavioural Intervention for Tics (ORBIT) randomized controlled trial for children and young people. Trials. 2020 Jan 2;21(1):6. doi: 10.1186/s13063-019-3974-3. PMID 31898510
- [Derived] Hall CL, Davies EB, Andren P, Murphy T, Bennett S, Brown BJ, Brown S, Chamberlain L, Craven MP, Evans A, Glazebrook C, Heyman I, Hunter R, Jones R, Kilgariff J, Marston L, Mataix-Cols D, Murray E, Sanderson C, Serlachius E, Hollis C; ORBIT Trial team.. Investigating a therapist-guided, parent-assisted remote digital behavioural intervention for tics in children and adolescents-'Online Remote Behavioural Intervention for Tics' (ORBIT) trial: protocol of an internal pilot study and single-blind randomised controlled trial. BMJ Open. 2019 Jan 3;9(1):e027583. doi: 10.1136/bmjopen-2018-027583. PMID 30610027